CLINICAL TRIAL: NCT05111938
Title: Friends, Family and Food: Interactive Virtual Environments for Children With Food Allergies - II
Brief Title: Friends, Family & Food: Food Allergy App for Youth - II
Acronym: F3A-App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Virtually Better, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: R42 HD075524 (RCT); R42HD075524 (NIH)
Record Dates: First submitted 2021-10-07; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-05

CONDITIONS: Food Allergy in Children
Keywords: food allergy; intervention; virtual; pediatric
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: AB/BA crossover: participants were randomized to Arm A (Standard Care (SC) then F3A-App), or Arm B (F3A-App then SC)
Who Masked: Outcomes Assessor
Masking Description: Research assistants were masked to treatment condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Standard Care followed by F3A-App (Active Comparator): The first portion of Arm A is a Standard Care (SC) office visit. Changes over time in Arm A represent a typical delivery channel in which a physician provides brief education and then encourages use of the F3A-App program. The SC intervention included a brief, structured office visit designed to replicate what would typically occur in a follow-up visit in an allergy clinic, and include provision standardized educational handouts available from the Food Allergy Research & Education (FARE) website. The second phase of Arm A is use of the F3A-App.
  Interventions: Behavioral: Friends, Family, and Food App (F3A-App)
- Arm B: F3A-App followed by Standard Care (Active Comparator): The first portion of Arm B is the use of the F3A-App for 2 weeks. Changes over time in Arm B represent an alternative delivery channel in which families use the F3A-App on their own and then have a follow-up office visit after using the self-guided program. The second phase of Arm B is the standard care office visit.
  F3A-App efficacy vs. SC is evaluated after the first intervention period on primary outcomes.
  Interventions: Behavioral: Friends, Family, and Food App (F3A-App)

INTERVENTIONS:
Behavioral: Friends, Family, and Food App (F3A-App)

SUMMARY:
Objective: This Phase II STTR grant incorporated user feedback collected in an earlier development project to build interactive, web-based software that helps children with food allergies learn about their condition and gain self-management skills. This highly interactive game allows children to progress through virtual scenes to help them learn about food avoidance, symptom detection, and reaction management. In addition, this project built gaming complexity, with more levels and game options, of the two interactive games "Label Learning: Like it or Lose it!" and "Reaction Action!." Research Procedures: The researchers elicited input from 8 families of children (ages 8-12) with food allergies and their parents by presenting some of preliminary intervention materials (e.g., storyboards of a child in a family gathering involving food) in a focus group format. After that, up to 40 families of children with food allergies (ages 8-12) were recruited to participate in an "open trial". Families were asked to use the software for two weeks and provide feedback on the software. Up to 100 families of children with food allergies (ages 8-12) were then recruited to participate in a Randomized Clinical Trial (RCT) to assess the efficacy of the F3A-App vs. Standard Care (brief office visit and educational handouts). Families in the clinical trial were asked to use the software for two weeks and complete a standard care allergy office visit. This design enabled the investigators to evaluate combined effects of Standard Care and the F3A-App through typical treatment channels (e.g., is the greatest efficacy found after a physician refers family to use the App after an office visit?). Gains in families' knowledge and confidence in food allergy management were evaluated, and interviews with families were conducted to gain further input regarding the software's credibility, usability, and acceptability.

This entry describes only the RCT portion of this Phase II STTR project.

DETAILED DESCRIPTION:
The central goal of this project was to develop an interactive, game-based application (App) for school-aged children (aged 8-12) with food allergies (FA) that would increase knowledge, improve behavioral skills for disease management, and ultimately reduce risk of negative outcomes. An effective FA intervention for children should target content areas of food avoidance and reaction management, and across these areas facilitate knowledge acquisition, develop behavioral skills, and provide practice using these skills in social contexts. The "Friends, Family, and Food App (F3A-App)", consists of four related parts: (a) an interactive, game-based application that is the core of the program, (b) the experiential scenarios in interactive environments (e.g., school cafeteria vignette) that target knowledge and behavioral skills practice in social contexts, (c) two engaging multi-level games to build skills in food avoidance (Label Learning: Like it or Lose it!) and symptom assessment (Reaction Action!), and (d) a multi-tiered reward system that uses token economy-based reinforcement to enhance motivation and engagement (SeaLife Spectacular). From a user perspective, the interactive, game-based application provides opportunities to practice behavioral skills (e.g. negotiating pressures to accept trigger foods, requesting assistance from adults, responding to teasing/bullying) in role-play situations with immediate feedback and reinforcement.

In this Phase II project, the investigators proposed to produce a fully-developed version of the F3A-App, including added content and enhanced features, and evaluate the final product in a randomized clinical trial.

The specific aims of Phase II were:

1. To refine the F3A-App based on the user feedback and data collected in Phase I.
2. To develop and field test additional content, including two additional interactive environments (family gathering, school pot-luck); and to increase gaming complexity (i.e., more levels and options) in Label Learning: Like it or Lose it! and Reaction Action! A small open trial was conducted, in which 40 children with FA, ages 8-12, used selected segments containing the newly developed content. Children used the application for 2 weeks on their home computer or tablet. Feedback about device preference and usage was used to determine the focus of the Evaluation Stage (Aim 3).
3. To assess the efficacy of the F3A-App vs. Standard Care (brief office visit and educational handouts) in a randomized clinical trial with 100 children with FA, ages 8-12. The investigators expected the F3A-App would improve children's FA knowledge and self-efficacy to manage FA (primary outcomes) and would increase parent-child communication regarding FA management relative to Standard Care (secondary outcome). The study's crossover design also made it possible to evaluate combined effects of Standard Care and the F3A-App through typical treatment channels (e.g., is the greatest efficacy found after a physician refers family to use the App after an office visit?) This Phase II STTR targeted pediatric FA, a critical public health problem of increasing prevalence. The approach was innovative by incorporating an emphasis on behavioral skills practice using a platform that is engaging, interactive, affordable, and has high potential for broad dissemination. The researchers envision that the F3A-App will ultimately serve as a template for interactive, game-based applications for children with other chronic conditions requiring self-management, such as asthma, diabetes, and celiac disease.

This entry describes only the RCT portion of this Phase II STTR project.

ELIGIBILITY:
Inclusion Criteria:

1. child must be 8-12
2. child must have an active diagnosis of FA, confirmed by a physician
3. child and parent must speak and read English
4. child must have access to a computer with internet access
5. child must have access to a smartphone or table

Exclusion Criteria:

any chronic health condition requiring substantial dietary self-management (e.g., diabetes)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Change in Food Allergy Management Assessment Scale (FAMAS) scores | Change in various elements of FA management (pre/post F3A-App use or Standard Care office visit, depending on randomized group assignment)
  Semi-structured interview assessing various elements of food allergy (FA) management (caregiver and youth report). Domains of the scale are: FA knowledge, symptom assessment, family/child response to allergic reactions, family/child food avoidance, medication availability, alternate caregivers, parent/child anxiety related to FA, balanced integration of FA and family life. Higher scores on all scales indicate more optimal FA management. Klinnert, M.D., et al., Children's food allergies (FA): Development of the Food Allergy Management and Adaptation Scale (FAMAS). Journal of Allergy and Clinical Immunology, 2012. 129(AB299).
Change in scores on the Food Allergy Independent Measure (FAIM) | Change in FA-related anxiety (pre/post F3A-App use or Standard Care office visit, depending on randomized group assignment)
  The FAIM is a 4-item measure of anxiety related to the child's food allergy. Higher scores indicate a higher degree of anxiety. van der Velde J. L., Flokstra-de Blok B. M. J., Vlieg-Boerstra B. J., Oude Elberink G., DunnGalvin A., Hourihane J. B., Dubois A. E. J. (2010). Development validity and reliability of food allergy independent measure (FAIM). Allergy, 65, 630-635. doi: 10.1111/j.1398-9995.2009.02216.x
Change in scores on the Food Allergy Self-Efficacy | Change in self-efficacy related to self-tx of FA (pre/post F3A-App use or Standard Care office visit, depending on randomized group assignment)
  Self-efficacy related to self-treatment of Food Allergy (youth report). Higher scores indicate a higher level of self-efficacy. Bursch, B., et al., Construction and validation of four childhood asthma self-management scales: parent barriers, child and parent self-efficacy, and parent belief in treatment efficacy. J Asthma, 1999. 36(1): p. 115-28.
Change in Food Allergy Knowledge scores | Change in FA-related knowledge (pre/post F3A-App use or Standard Care office visit, depending on randomized group assignment)
  An assessment of the level of food allergy-related knowledge (youth report). Higher scores indicate better knowledge of FA. Sicherer, S.H., et al., Development and validation of educational materials for food allergy. Journal of Pediatrics, 2012. 160(4): p. 651-656.
Change in Parent-Child Communication related to Food Allergy | Change in amount of parent-child discussion related to FA (pre/post F3A-App use or Standard Care office visit, depending on randomized group assignment)
  This measure was adapted from a parent-child communication assessment used to evaluate communication about sexual health. The Food Allergy adaptation evaluates the number of times parent and child discussed each of 6 FA management topics in prior week (e.g., using epinephrine) (caregiver and youth report). Huston, R.L. and L.J. Martin, Effect of a program to facilitate parent-chld communication about sex. Clinical Pediatrics, 1990. 29(11): p. 626-633.
  45. Schuster, M.A., et al., Evaluation of talking parents, healthy teens, a new worksite based parenting programme to promote parent-adolescent communication about sexual health: randomised controlled data. BMJ, 2008. 337(a308).

OTHER OUTCOMES:
Acceptability of the Friends, Family and Food App (F3-App): Technology Post-Trial Impressions Questionnaire | Follow up (after use of the F3-App; approximately 8 week after baseline)
  Standard user experience questions were adapted to elicit feedback from study participants regarding the logic of F3-App, participants' confidence in their FA treatment, and whether they would recommend the F3-App to others. Borkovec, T. D., & Nau, S. D. (1972). Credibility of analogue therapy rationales. . Journal of Behavior Therapy & Experimental Psychiatry, 3, 257-260. 31. Silverman, W. K., Kurtines, W. M., Ginsburg, G. S., Weems, C. F., Lumpkin, P. W., & Carmichael, D. H.
  (1999). Treating anxiety disorders in children with group cognitive-behaviorial therapy: a randomized clinical trial. J Consult Clin Psychol, 67(6), 995-1003. 32. Witmer, B. G., & Singer, M. J. (1998). Measuring Presence in Virtual Environments: A Presence Questionnaire. Presence: Teleoperators and Virtual Environments, 7(3), 225-240.
Credibility of the F3-App: Technology Post-Trial Impressions Questionnaire | Follow up (after use of the F3-App; approximately 8 week after baseline)
  Degree of realism (visuals, audio) and participants' game interest were evaluated using items adapted from standard user experience measures. Borkovec, T. D., & Nau, S. D. (1972). Credibility of analogue therapy rationales. . Journal of Behavior Therapy & Experimental Psychiatry, 3, 257-260. 31. Silverman, W. K., Kurtines, W. M., Ginsburg, G. S., Weems, C. F., Lumpkin, P. W., & Carmichael, D. H.
  (1999). Treating anxiety disorders in children with group cognitive-behaviorial therapy: a randomized clinical trial. J Consult Clin Psychol, 67(6), 995-1003. 32. Witmer, B. G., & Singer, M. J. (1998). Measuring Presence in Virtual Environments: A Presence Questionnaire. Presence: Teleoperators and Virtual Environments, 7(3), 225-240.
Adherence to the use of the F3-App during study | Follow up (after use of the F3-App; approximately 8 week after baseline)
  Percentage of completed modules & games
Food Allergy Caregiver-Child Communication | Baseline and Follow up (after use of the F3-App; approximately 8 week after baseline)
  Caregiver & Child report versions. Eight yes/no questions about topics discussed between caregiver and child in previous week.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Mann-Koepke, PhD, Study Chair — Eunice Kennedy Shriver National Institute of Child Health & Human Development (NICHD)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jandasek BN, Kopel SJ, Esteban CA, Rudders SA, Spitalnick JS, Larsen MA, Cushman GK, McQuaid EL. Friends, Family, and Food: Development of a Food Allergy Intervention, F3-App, for Children. Clin Pract Pediatr Psychol. 2024 Jun;12(2):143-156. doi: 10.1037/cpp0000513. Epub 2024 Jan 8. PMID 39045229